CLINICAL TRIAL: NCT06327113
Title: A Phase 2 Randomized Study Comparing Subcutaneous Tumescent Antibiotic Administration With Standard of Care for the Treatment of Chronic Wounds
Brief Title: Antibiotic Tumescent For Chronic Wounds
Acronym: TAI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Seth J Putterman, Professor of Physics and Astronomy at University of California, Los Angeles, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#23-001248
Record Dates: First submitted 2024-02-28; First posted 2024-03-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Non-healing Wound
Keywords: chronic wound; wound care
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: This is a single center, prospective, comparative interventional, two-arm parallel group, randomized, clinical safety and efficacy trial comparing a group receiving standard wound care with tumescent antibiotic injection (TAI) with a control group receiving standard wound care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Wound Care) (No Intervention): The 'control' group will receive wound care treatment in accordance to standard of care procedures. The 'control' group will not receive study intervention.
- Treatment Group (Tumescent Antibiotic Injection) (Experimental): The 'treatment' group will receive wound care treatment in accordance to standard of care procedures along with the study intervention, a one-time tumescent antibiotic injection (TAI).
  Interventions: Drug: CeFAZolin Injectable Solution

INTERVENTIONS:
Drug: CeFAZolin Injectable Solution — One gram Cefazolin reconstituted in 100 mL 0.9% Sodium Chloride (normal saline)
  Other Names: Kefzol, Ancef
  Arms: Treatment Group (Tumescent Antibiotic Injection)

SUMMARY:
Chronic non-healing wounds are becoming an increasingly more common problem. Eligible, consenting patients with chronic wounds in the lower extremities, upper extremities or trunk, will either continue to the standard of care or will be randomized to the treatment cohort where antibiotic solution will be injected in the area around the wound. All patients will continue standard wound care as dictated by the wound care clinic. Subjects of both the control and treatment will have approximately 6 study specific visits that may or may not coincide with previously schedule wound care clinic visits. As these specified visits wound size and healing will be documented and patients will complete surveys. The study will conclude for the subject after approximately 6 months. Again, these patients may continue standard wound care but will no longer have study obligations.

DETAILED DESCRIPTION:
Foot ulcers develop in 9.1-26 million people with diabetes annually worldwide. Up to 1% of people in industrialized countries will suffer from a leg ulcer. Numbers of pressure and venous ulcers are rising at rates of 6-7% annually, diabetic ulcers rising at 9%. In the United States, chronic wounds affect 6.5 million patients and over $25 billion dollars are spent annually on chronic wound care. Medicare spending on pressure and arterial ulcers in 2014 was $3696 and $9015 per patient. Diabetic limb complications are more costly than breast cancer.

Attempts to treat chronic wounds have included 1) debridement, 2) specialized dressings, 3) compression bandages, 4) negative pressure devices, 5) topical growth factors and pharmaceuticals, 6) skin grafts and skin substitutes, 7) hyperbaric oxygen therapy and 8) amputation. There is no study that examines the utility of tumescent antibiotic injections (TAI) into a wound. TAI is a relatively simple, cost-effective procedure using known, drugs with a well characterized safety profile, and used in a new way to address this large unmet need.

Our group has published work in this area showing appropriate design, feasibility and safety in a large animal model. The investigators have shown that direct antibiotic delivery through tumescent injections can achieve high antibiotic concentrations directly in skin and soft tissue for sufficient time to kill bacteria. Simultaneously, total antibiotic doses can be kept low, minimizing systemic toxicity. In particular, even antibiotic resistant strains of pathogenic microorganisms may be susceptible due to the high local concentration of antimicrobial agent. Tumescent injections can more effectively deliver antibiotic to compromised body regions with impaired circulation compared to intramuscular or intravenous drug delivery.

Primary Objective

1. To assess the safety of tumescent antibiotic injections.

Secondary Objectives

1. To evaluate wound size or closure.
2. To evaluate chronic-wound-related pain.
3. To evaluate Quality of Life.

Exploratory Objectives

1. Assess the number of chronic wound-related complications (increased wound sizes, infections, dermatitis).
2. Assess the number of clinical signs of infection in participants.
3. Determine the species of pathogenic bacteria present in wound.

Screening: up to 1 week. Treatment: TAI will take 1 day. Standard wound care will be ongoing until the wound closes, as it would in a wound care center.

Follow-up:

Once weekly (+/-1 week) for 2 weeks, followed by Biweekly (+/-1week) for 4 more weeks. There will also be a 3 month (+/- 2 weeks) and 6 month (+/- 4 weeks) follow up visits. Total duration of participant participation is up to approximately 1 year. Total duration of the study for recruitment and completion of visits is expected to be up to two years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Must have:

  1. One or more full thickness ulcers on the lower extremity, upper extremity (excluding the hands) or trunk with a surface area exceeding 0.5 cm^2 (50 mm^2) and less than 30 cm^2 (6*5 cm) after debridement (full thickness means extending through the epidermis and dermis but not involving tendon, bone or joint capsule).
  2. Presence of a chronic wound (including venous ulcer, arterial ulcer, below knee pressure ulcer, diabetic foot ulcer, ischemic ulcer) that has existed for >4 weeks at Visit 1.
  3. Documentation that the wound has been treated at least 2 times at the wound care center.
  4. Documentation that the wound area has not decreased by more than 50% in 4 weeks.
  5. Willing to provide written informed consent (and assent when applicable) obtained from participant or participant's legal representative and ability for participant to comply with the requirements of the study.
* Adequate perfusion as demonstrated by TcPO2≥40 mm Hg, ABI ≥ 0.7, or great toe pressure≥50 mm Hg, or palpable pulses of the lower extremity such as dorsalis pedis and/or posterior tibial artery or palpable radial artery in the upper extremity.
* In the opinion of the investigator, participants must be considered reliable, willing, and able to give signed informed consent in English and sign the informed consent form.
* For participants of reproductive potential, two of the following forms of contraception are required between visits 1-4 (total of 3-6 weeks), one of which must be a barrier method:

  1. Condoms (male or female) with or without a spermicidal agent
  2. Diaphragm or cervical cap with spermicide
  3. Intrauterine device (IUD)
  4. Tubal ligation
  5. Hormone-based contraceptive such as oral birth control pills

Exclusion Criteria:

* Participants with limb threatening infection, extensive cellulitis (≥2 cm radially beyond the borders of the wound), lymphangitis, fasciitis, deep tissue infection, abscess, pus, osteomyelitis, or other evidence of local or systemic complications of infection.

  1. Wound size/surface area, duration, severity, or location outside of INCLUSION criteria Note: Consideration will be given to minor variation, if deemed appropriate by the medical director, and authorized.
  2. Clinically severe wound at high risk for amputation as determined by the Medical Director.
  3. All pressure ulcers except below knee pressure ulcers.
* Cellulitis or acute infection as determined by:

  1. Significant wound erythema, induration, warmth, presence of pus, or tenderness, determined by PI or medical director ≥ 2 cm radially from wound margin.
  2. Fever with electronic temp >100.4°F (>38°C)
* Following enrollment, if wound culture returns positive for Pseudomonas.
* Participants with symptoms of systemic infection or uncontrolled diabetes mellitus (e.g., severe hyperglycemia, ketoacidosis, azotemia).
* Participants who are allergic or have shown hypersensitivity to penicillin, cefazolin, other beta-lactams, the cephalosporin group of antibiotics, lidocaine, or to local anesthetics of the amide type.
* Participants requiring intravenous antimicrobials during the study period for any infection, including diabetic foot ulcer. Mild localized infection that would be treated on an outpatient basis could be approved by Medical Director authorization.
* Participants who are currently treated by dialysis, awaiting dialysis, or who have an estimated glomerular filtration rate of ≤ 30 mL/min/1.73 m^2.
* Participants who are expected to be unable to care for their ulcer because of hospitalization, vacation, disability, etc., during the study period.
* Participants with known active alcohol or substance abuse within the 6 months preceding study entry.
* Participants who are receiving systemic corticosteroids (in a dose equivalent to ≥20 mg of prednisone per day), biologic therapy, immunosuppressants, , radiation therapy, or cytotoxic agents, unless approved by medical director authorization
* Participants who require treatment for a primary or metastatic malignancy (other than squamous or basal cell carcinoma of the skin, not involving the wound site).
* Participants with acquired immune deficiency syndrome (AIDS) or known human immunodeficiency virus (HIV) positivity.
* Participants with other conditions considered by the investigator to be reasons for disqualification that may jeopardize participant safety or interfere with the objectives of the trial (e.g., acute illness or exacerbation of chronic illness, lack of motivation, history of poor compliance).
* Women who are breastfeeding, pregnant, or attempting to become pregnant.
* Active acute medically unstable condition defined by:

  1. Diabetes Mellitus Type 1 or 2, with A1C greater than 9.5. Consideration to HbA1c higher than 9.5 - 10.0% after consultation with the medical director or PI.
  2. Unstable cardiovascular or other high-risk general medical condition making participation in the study a significant risk to the participant, per medical director determination.
  3. Laboratory evidence of severe metabolic, renal, hepatic, endocrine, hematologic disorder per medical director determination.
  4. Recent trauma complicated by significant bone, nerve, or vascular damage.
  5. Sickle Cell Disease.
* Participant is enrolled/participating in another study or does not agree to refrain from participating in another study while enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
Primary Objective - Assess the rate of occurrence and severity of adverse events and their relationship to TAI | From enrollment through 6 month visit.
  Adverse events will be tabulated by treatment group and will include the number of participants for whom the event occurred, the rate of occurrence, and the relationship to TAI. The severity of adverse events will be measured by the adverse event severity scale (1-4; Mild; Moderate; Severe; Life-threatening). The relationship of the adverse event to the study drug will be assessed by the likelihood of the relationship (Definitely; Probably; Possibly; Unrelated). Frequency of adverse events that result in discontinuation of the investigative treatment will be quantified.

SECONDARY OUTCOMES:
Secondary Objective - To evaluate wound size and closure. | From enrollment through 6 month visit or until wound is closed.
  Wound closure will be determined by the clinical practitioner at time of wound assessment at clinic follow up. If wound is not closed, wound size will be measured with a device that scans the wound and determines its area in cm^2. If wound is closed the wound size will be returned as 0 cm^2.
Secondary Objective - Chronic-wound-related pain | From enrollment through 6 month visit.
  Chronic wound-related pain will me be measured with a pain assessment administered every visit. The pain assessment is the PEG-3 Pain Screening Tool which consists of 3 questions; The PEG-3 answer scale ranges from 0 to 10 for each question, where 0 corresponds to no pain and 10 represents the worst pain. A combined score is generated by summing the answer to each question.
Secondary Objective - Rating Quality of life | From enrollment through 6 month visit.
  Quality of Life (QoL) will be measured with a QoL assessment administered at every visit.
  The QoL assessment is the WOUND-QOL-14 QUESTIONNAIRE which consists of 14 questions. Answers to each item are coded with numbers (0='not at all', 1='a little', 2='moderately', 3='quite a lot', to 4='very much') and summed or averaged to generate a global score. A higher score denotes a lower QoL.

OTHER OUTCOMES:
Exploratory Objectives - Assess the number of chronic wound-related complications (increased wound sizes, infections, dermatitis). | From enrollment through 6 month visit.
  Record the number and severity of chronic-wound-related complications.
  1. difference in wound size,
  2. incidence and degree of infection
  3. occurrence of dermatitis.
  4. Difference in wound quality via visual inspection (granulation tissue, tissue necrosis, exudate, drainage).
Exploratory Objectives - Assess the number of clinical signs of infection in participants. | From enrollment through 6 month visit.
  Record number and severity of clinical signs of infection.
  1. cellulitis via visual inspection and exam,
  2. pus via visual inspection and exam,
  3. fever via visual inspection and exam,
  4. abscess via visual inspection and exam.
Exploratory Objectives - Determine the species of pathogenic bacteria present in wound. | From enrollment through 6 month visit.
  Species of pathogenic bacteria will be determined with a wound culture.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Putterman, PhD, Study Director — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] O'Meara S, Cullum N, Nelson EA, Dumville JC. Compression for venous leg ulcers. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD000265. doi: 10.1002/14651858.CD000265.pub3. PMID 23152202
- [Background] Krzyszczyk P, Schloss R, Palmer A, Berthiaume F. The Role of Macrophages in Acute and Chronic Wound Healing and Interventions to Promote Pro-wound Healing Phenotypes. Front Physiol. 2018 May 1;9:419. doi: 10.3389/fphys.2018.00419. eCollection 2018. PMID 29765329
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Nussbaum SR, Carter MJ, Fife CE, DaVanzo J, Haught R, Nusgart M, Cartwright D. An Economic Evaluation of the Impact, Cost, and Medicare Policy Implications of Chronic Nonhealing Wounds. Value Health. 2018 Jan;21(1):27-32. doi: 10.1016/j.jval.2017.07.007. Epub 2017 Sep 19. PMID 29304937
- [Background] Barshes NR, Sigireddi M, Wrobel JS, Mahankali A, Robbins JM, Kougias P, Armstrong DG. The system of care for the diabetic foot: objectives, outcomes, and opportunities. Diabet Foot Ankle. 2013 Oct 10;4. doi: 10.3402/dfa.v4i0.21847. PMID 24130936
- [Background] Koulakis JP, Rouch J, Huynh N, Wu HH, Dunn JCY, Putterman S. Tumescent Injections in Subcutaneous Pig Tissue Disperse Fluids Volumetrically and Maintain Elevated Local Concentrations of Additives for Several Hours, Suggesting a Treatment for Drug Resistant Wounds. Pharm Res. 2020 Feb 10;37(3):51. doi: 10.1007/s11095-020-2769-2. PMID 32043171
- [Background] Nicolau DP, Silberg BN. Cefazolin potency against methicillin-resistant Staphylococcus aureus: a microbiologic assessment in support of a novel drug delivery system for skin and skin structure infections. Infect Drug Resist. 2017 Jul 26;10:227-230. doi: 10.2147/IDR.S134497. eCollection 2017. PMID 28794647
- [Background] Okuma K, Iwakawa K, Turnidge JD, Grubb WB, Bell JM, O'Brien FG, Coombs GW, Pearman JW, Tenover FC, Kapi M, Tiensasitorn C, Ito T, Hiramatsu K. Dissemination of new methicillin-resistant Staphylococcus aureus clones in the community. J Clin Microbiol. 2002 Nov;40(11):4289-94. doi: 10.1128/JCM.40.11.4289-4294.2002. PMID 12409412
- [Background] Durand BARN, Pouget C, Magnan C, Molle V, Lavigne JP, Dunyach-Remy C. Bacterial Interactions in the Context of Chronic Wound Biofilm: A Review. Microorganisms. 2022 Jul 25;10(8):1500. doi: 10.3390/microorganisms10081500. PMID 35893558
- [Background] Kim H, Park H, Lee SJ. Effective method for drug injection into subcutaneous tissue. Sci Rep. 2017 Aug 29;7(1):9613. doi: 10.1038/s41598-017-10110-w. PMID 28852051
- [Background] Scali C, Kunimoto B. An update on chronic wounds and the role of biofilms. J Cutan Med Surg. 2013 Nov-Dec;17(6):371-6. doi: 10.2310/7750.2013.12129. PMID 24138971
- [Background] Boeni R. Safety of tumescent liposuction under local anesthesia in a series of 4,380 patients. Dermatology. 2011;222(3):278-81. doi: 10.1159/000327375. Epub 2011 May 24. PMID 21606638
- [Background] Harb G, Lebel F, Battikha J, Thackara JW. Safety and pharmacokinetics of subcutaneous ceftriaxone administered with or without recombinant human hyaluronidase (rHuPH20) versus intravenous ceftriaxone administration in adult volunteers. Curr Med Res Opin. 2010 Feb;26(2):279-88. doi: 10.1185/03007990903432900. PMID 19947907
- [Background] Coerper S, Beckert S, Kuper MA, Jekov M, Konigsrainer A. Fifty percent area reduction after 4 weeks of treatment is a reliable indicator for healing--analysis of a single-center cohort of 704 diabetic patients. J Diabetes Complications. 2009 Jan-Feb;23(1):49-53. doi: 10.1016/j.jdiacomp.2008.02.001. Epub 2008 Apr 3. PMID 18394932
- See also: UCLA Center for Wound Healing & Limb Preservation — https://www.uclahealth.org/locations/ucla-center-wound-healing-limb-preservation